

# MUHIMBILI UNIVERSITY OF HEALTH AND ALLIED SCIENCES (MUHAS)

Title: Entrepreneurship and Beekeeping for Young Men at Risk for Violence: a pilot study2014-

ID: 11-07/AEC/Vol.IX/35

Consent Form

Date: December 2014



Consent Form Date: December 2014

Title: Entrepreneurship and Beekeeping for Young Men at risk for Violence, Tanzania: Piloting an Intervention

Sponsor: Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

Principle Investigator:

Address: School of Nursing, PO Box 65004, Dar es Salaam, Tanzania

### Introduction

This consent form contains information about the research named above. In order to be sure that you are informed about being in this research, we are asking you to read (or have read to you) this consent form. You will also be asked to sign it (or make your mark in front of a witness). We will give you a copy of this form. This consent form might contain some words that are unfamiliar to you. Please ask us to explain anything you may not understand.

#### Reason for the Research

You are being asked to take part in research to help us to learn how to decrease violence in Dar es Salaam and how to develop effective interventions.

# General Information about Methods

If you agree to this research, you will be interviewed. We will ask you questions about your socio-economic background, health, economic needs, and your aspirations for the future. You will be take part in training sessions on health and/or economic empowerment and/or beekeeping. We will then interview you three more times, after the training sessions are complete.

# Your part in the research

If you agree to be in the research, you will be asked questions from the pre-tested questionnaire. You will agree to participate in 2-10 training sessions, each training session will last for one day. About fifty youth will take part in this research which is being conducted at the Kibaha Beekeeping Training Center.

#### Possible risks

This research will ask you questions that you may find sensitive, touching some aspects of your life. You may feel free to choose not to answer any questions that you don't feel like answering. If you are working with bees, it is possible you could be stung by a bee. You will be taught how to handle bees carefully, and a nurse will be near by to administer first aid if necessary.

#### Possible benefits

What we learn from you will be useful for this country and the world as well. The findings of this study will help in establishing effective work oriented interventions for youth. In addition you will receive training in health, and/or economic empowerment, and/or beekeeping that will aid you in your life.

If you decide not to be in this research

You are free to decide if you want to be in this research.

#### Confidentiality

We will protect information about you and your taking part in this research to the best of our ability. You will not be named in any reports. However the principle investigators may sometimes look at your research records. You do not have to answer questions that you do not want. You may also ask for clarification of some questions that you do not understand. In the future we will want to interview you again, so we expect to make follow up. We may contact you by phone or in person at the camp to see if you still want to take part in the research.

# Compensation

You will be compensated for your bus fare to reach training sessions. You will receive lunch on days of official training sessions, and a small per diem to compensate for your time.

# Leaving the Research

You may leave the research at any time. If you choose to take part, you can change your mind at any time and withdraw.

If so, please tell the researchers why you wish to leave.

Also, you may be asked to leave the research if:

- the research staff feel it is best for you
- if you react strongly to a bee sting
- the research is stopped.

| If you have a Problem or Other Questions | |
|---|---|
| If you have a problem that you think might be related to taking part in this research or any | |
| questions about the research please call | , mobile phone number |
| If you need more help, we may advice for further evaluation or referral. | |

Your Rights as a Participant

This research has been reviewed and approved by the Research and Publications Directorate of Muhimbili University of Health and Allied Sciences. This is the committee that reviews research studies in order to help protect participants. If you have any questions about your rights as a research participant, you may contact Dr. JRP Masalu, phone number 255 22 2152489, PO Box 65001, Dar es Salaam, Tanzania.

# Volunteer Agreement

The above document describing the benefits, risks, and procedures for the research titled: Youth Unemployment, Community Violence, and Creating Opportunities: Piloting an Intervention, RukaJuu Beekeeping has been read and explained to me. I have been given an oppiortunity to have any questions about the research answered to my satisfaction. I agree to participate in this research

Date

Signature or thumb print

If participants cannot read the form themselves, a witness must sign here: I was present while the benefits, risk and procedures were read to the potential participant. All questions were answered and the potential participant has agreed to take part in the research.

Date

Signature of Witness